CLINICAL TRIAL: NCT04351425
Title: Feasibility and Safety of Earlier Weaning of Preterm Newborn From Incubator to Cot at 1400 Grams
Brief Title: Early Weaning of Preterm Newborn From Incubator to Cot at 1400 Grams
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Abdulrahman Al-Matary, Principal Investigator, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-048
Record Dates: First submitted 2019-09-18; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Pre-Term; Body Temperature Changes; Transition; Patient Discharge; Length of Stay
Keywords: Preterm; Patient discharge; Length of stay; Low birth weight
MeSH Terms: conditions — Premature Birth; Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: This was a randomized control trial with preterm neonates with birth weights < 1400 g conducted at King Fahad Medical City, Riyadh, Saudi Arabia. We compared newborns weaned to cot at a weight of 1400 g to newborns weaned at a weight of 1600 g. The outcome was to assess the feasibility of the protocol in terms of temperature control and average weight gain.
Masking Description: Participants: randomly selected infants, group 1 less than 1400 kg, group 2 more than 1600 kg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- study group (Experimental): study group will be shifted from incubator to an unheated open cot a weight of 1400 grams
  Interventions: Device: Weaning to crib; Device: Weaning from incubator
- control group (Active Comparator): control group will be shifted from incubator to an unheated open cot at a weight of 1600 grams
  Interventions: Device: Weaning to crib; Device: Weaning from incubator

INTERVENTIONS:
Device: Weaning to crib — We weaned the infants into two groups. Group A, 1.6 kg
  Other Names: Giraffe GELV61778 General Electric Company
Device: Weaning from incubator — We weaned the infants into two groups. group B, 1.4 kg
  Other Names: Giraffe GELV61778 General Electric Company

SUMMARY:
Background: To maintain the body temperature of preterm newborns is one of the essential criteria for discharge from hospital.

Aim: we aimed to assess the feasibility and the safety of an early weaning protocol from incubator to unheated cot at 1400 g preterm newborns.

Methods: This was a randomized control trial with preterm neonates with birth weights < 1400 g conducted at King Fahad Medical City, Riyadh, Saudi Arabia. We compared newborns weaned to cot at a weight of 1400 g to newborns weaned at a weight of 1600 g. The outcome was to assess the feasibility of the protocol in terms of temperature control and average weight gain.

Results: A total of 23 preterm neonates were recruited in this study. The baseline characteristics were similar except for the gestational age was higher in the newborns enrolled to 1400 g group. Early weaning was achieved in 100% of newborns without significant adverse effects on temperature stability or weight gain. Incidence of low and high temperatures per newborn and the average weight gain before and after transfer and after transfer were not different between the two groups.

Conclusion: Our results showed the feasibility and safety of 1400 g weaning protocol for preterm newborns, without any adverse effects or increasing the neonatal length of hospital stay. Further investigations in larger patient groups are recommended.

DETAILED DESCRIPTION:
1. Introduction To discharge a preterm newborn after staying in neonatal intensive care unit (NICU) is a multifactorial decision. According to the American Academy of pediatrics guidelines of the physiologic competencies for hospital discharge of the high-risk neonate including preterm ones, are sufficient oral feeding and mature respiratory control, and finally the ability to maintain a normal body temperature in an unheated open bed (1). These mostly are achieved between 36 and 37 weeks' postmenstrual age (2-4).

   Shortening the period of a hospital stay, it could be beneficial to decrease the emotional stress resulted from the separation between the mother and the newborn and parents; furthermore, it may reduce the hospital-acquired co-morbidities as sepsis and surgical needs (5) and accordingly reduce the economic burden on the society.

   The timing to wean from the incubator is crucial since the immaturity of preterm newborn's thermoregulatory mechanisms which could affect weight gain as an attempt to maintain body temperature, achieving full feeding volume, and as a result could delay discharge from hospital (6, 7). The target weight for incubator weaning varies widely among NICUs. The common usual practice is between of 1700-1800 g, and it is generally based on the professional experience and judgment (8, 9).

   In 2010, a Cochrane Review assessed transferring preterm infants from incubator to open bed at a lower body weight (˂1700 g) by comparing to a higher body weight (˃ 1700 g). The review showed that preterm newborns can be transferred to open beds at 1600 g without adverse effects on temperature stability in terms of return to incubator or daily weight gain (10). A multicenter trial achieved the same result (11).

   Moreover, there are few studies showed that infants can be successfully transferred into cots at weights down to 1500 g (9, 12). A pilot study carried out stepwise four cohort trials of newborn's transfer from incubators to open beds at 1800 g, then at 1700 g, then at 1600 g and then finally at 1500 g (13). It demonstrated that there were no significant differences between the four cohorts in maintain body temperature after incubator weaning.

   The primary outcome of this study was to evaluate the feasibility and safety of incubator weaning for medically stable preterm neonates to unheated open cot at a body weight of 1400 g in terms of daily weight gain and temperature control. Newborns in the same study period were compared to a control group weaned at body weight of 1600 g.
2. Subjects and Methods:

2.1. Study design A prospective randomized clinical trial was conducted at NICU at King Fahad Medical City, Riyadh, Saudi Arabia. Preterm newborns admitted to NICU fulfilling items in inclusion and exclusion criteria during the period from August 2017 to October 2018 were included into the study.

All eligible newborns were randomized into two groups to be weaned at 1,400 or at 1,600 g in a 1:1 ratio, using random block of 4. Newborns were eligible if body weight less than 1400 g, they were at least 5 days of age at the time of transferring to cot, they fed at least 60 ml/kg/day at the time of transferring to cot, and they are medically stable with no significant apnea or bradycardia, no ventilator support, no phototherapy and not having a major congenital abnormality. Newborns were excluded if they didn't fulfill the above criteria or unlikely to reach the target weight within 7 days.

2.2. Procedures Nursery temperatures were adjusted at 24-28 ◦c from birth to cot. The subjects were dressed in a hat, one vest and two wraps. Then, they were randomly assigned to either study group or control group. Infants were weighed naked daily. In the study group, the newborns were transferred to cot at a weight of 1400 to 1499 g and in the control group; they were transferred at a weight of 1600 to 1699 g. In the first day in the open cot, they were not bathed.

2.3. Data Collected

* Baseline characteristics as birth weight, gestational age (GA), gender, age in days in the transfer day, body weight and GA in the transfer day.
* Relevant data from to incubator weaning
* After transfer, hourly axillary temperatures were taken until two consecutive readings between 36.4 and 37.1 °C. Then, temperatures were taken every 3 hours with each feed for at least 72 hours. After that, temperatures were taken four times a day minimum until discharge. If the axillary temperature was ˂36.4°C, thus an additional wrap was added. If the temperature was still low for an hour later, then the infant was returned to the incubator. Meanwhile, if the temperature was more than 37.1°C, a wrap was reduced.
* No of infants who failed to be transferred to cot. Failure of transfer is defined as the inability to maintained body temperatures above 36.4°C in a two consecutive axillary temperatures in a cot despite of adding covering.
* For infants who remained in an open crib, the rate of weight gain calculated every day over the week before and after transfer. In the discharge day, age in days after transfer to discharge date, WT and GA.

2.4. Statistical methodology: Data were statistically described in terms of mean ± SD for continuous data and in frequencies (number of cases). For comparative purposes between groups in all continuous data, independent t-test or Mann Whitney t test was adopted. X2-square and fisher test were used for assessing association in categorical data.. P values less than 0.05 were considered statistically significant. All statistical calculations were done using computer program IBM SPSS (Statistical Package for the Social Science; IBM Corp, Armonk, NY, USA) release 21 for Microsoft Windows.

2.5. Ethical considerations: Due to safety concerns, the study was carried out in two steps. Initially, we started infants' weaning with the approved weaning weight at1500 grams. A total of 19 preterm infants were randomized in two groups. Both groups were weaned to cot with a 100% success rate without any complications. Afterwards, the study was approved by the local Ethics Committee to start the second phase of the study at weaning weight of 1400 g. The parents were all directly contacted and agreed in writing informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Clinical weight less than 1.5 kg at birth
* Clinically stable
* No cardio or respiratory support
* Reached 2/3 of his/her enteral feeding

Exclusion Criteria:

* IUGR
* Clinical unstable
* On cardio or respiratory support
* Dysmorphic

Ages: 23 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Estimated)
Dates: Start 2020-04-16 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
daily weight gain | 1 month
  newborns were weighed naked daily as a routine NICU practice using electronic scales. The rate of weight gain was calculated as grams/kilogram per day over the week before and after transfer.
temperature control | 1 month
  Hourly axillary temperature was taken until two consecutive readings of between 36.4 and 37.1 C, after which temperatures were taken 3 times with each feed until at least 72 hours after transfer and after that a minimum of four times a day until discharge. If the axillary temperature is less than 36.4◦C, an additional wrap was added. If the temperature remained low, an hour later, the newborn was returned to an incubator. Failure to transfer was defined as the inability to maintained body temperatures in a cot despite additional covering, with two consecutive axillary temperatures below 36.4 ◦C, one hour apart. If the temperature more than 37.1C°, the wraps were reduced accordingly.temperature

IPD SHARING:
Plan to Share IPD: No
If this study plan goes successfully through, we shall continue the study. Basically, there is no concern in regards to the safety of the participants

REFERENCES:
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn. Hospital discharge of the high-risk neonate. Pediatrics. 2008 Nov;122(5):1119-26. doi: 10.1542/peds.2008-2174. PMID 18977994
- [Background] Powell PJ, Powell CV, Hollis S, Robinson MJ. When will my baby go home? Arch Dis Child. 1992 Oct;67(10 Spec No):1214-6. doi: 10.1136/adc.67.10_spec_no.1214. PMID 1444564
- [Background] Brooten D, Kumar S, Brown LP, Butts P, Finkler SA, Bakewell-Sachs S, Gibbons A, Delivoria-Papadopoulos M. A randomized clinical trial of early hospital discharge and home follow-up of very-low-birth-weight infants. N Engl J Med. 1986 Oct 9;315(15):934-9. doi: 10.1056/NEJM198610093151505. PMID 3531852
- [Background] Casiro OG, McKenzie ME, McFadyen L, Shapiro C, Seshia MM, MacDonald N, Moffatt M, Cheang MS. Earlier discharge with community-based intervention for low birth weight infants: a randomized trial. Pediatrics. 1993 Jul;92(1):128-34. PMID 8390644
- [Background] Niknajad A, Ghojazadeh M, Sattarzadeh N, Bashar Hashemi F, Dezham Khoy Shahgholi F. Factors affecting the neonatal intensive care unit stay duration in very low birth weight premature infants. J Caring Sci. 2012 May 27;1(2):85-92. doi: 10.5681/jcs.2012.013. eCollection 2012 Jun. PMID 25276681
- [Background] Glass L, Silverman WA, Sinclair JC. Relationship of thermal environment and caloric intake to growth and resting metabolism in the late neonatal period. Biol Neonat. 1969;14(5):324-40. doi: 10.1159/000240198. No abstract available. PMID 4192368
- [Background] Gibson E, Medoff-Cooper B, Nuamah IF, Gerdes J, Kirkby S, Greenspan J. Accelerated discharge of low birth weight infants from neonatal intensive care: a randomized, controlled trial. The Early Discharge Study Group. J Perinatol. 1998 Nov-Dec;18(6 Pt 2 Su):S17-23. No abstract available. PMID 10023375
- [Background] New K, Bogossian F, East C, Davies MW. Practice variation in the transfer of premature infants from incubators to open cots in Australian and New Zealand neonatal nurseries: results of an electronic survey. Int J Nurs Stud. 2010 Jun;47(6):678-87. doi: 10.1016/j.ijnurstu.2009.10.017. Epub 2009 Nov 27. PMID 19945108
- [Background] Sutter TW, Phan D, Pierchala CE, Rishel W. Weaning of premature infants from the incubator to an open crib. J Perinatol. 1988 Summer;8(3):193-8. PMID 3225660
- [Background] New K, Flenady V, Davies MW. Transfer of preterm infants from incubator to open cot at lower versus higher body weight. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD004214. doi: 10.1002/14651858.CD004214.pub4. PMID 21901688
- [Background] Shankaran S, Bell EF, Laptook AR, Saha S, Newman NS, Kazzi SNJ, Barks J, Stoll BJ, Bara R, Gabrio J, Childs K, Das A, Higgins RD, Carlo WA, Sanchez PJ, Carlton DP, Pavageau L, Malcolm WF, D'Angio CT, Ohls RK, Poindexter BB, Sokol GM, Van Meurs KP, Colaizy TT, Khmour A, Puopolo KM, Garg M, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health, and Human Development Neonatal Research Network. Weaning of Moderately Preterm Infants from the Incubator to the Crib: A Randomized Clinical Trial. J Pediatr. 2019 Jan;204:96-102.e4. doi: 10.1016/j.jpeds.2018.08.079. Epub 2018 Oct 15. PMID 30337189
- [Background] Medoff-Cooper B. Transition of the preterm infant to an open crib. J Obstet Gynecol Neonatal Nurs. 1994 May;23(4):329-35. doi: 10.1111/j.1552-6909.1994.tb01884.x. PMID 8057186
- [Background] West CR, Williams M, Weston PJ. Feasibility and safety of early transfer of premature infants from incubators to cots: a pilot study. J Paediatr Child Health. 2005 Dec;41(12):659-62. doi: 10.1111/j.1440-1754.2005.00754.x. PMID 16398870
- [Background] Zecca E, Corsello M, Priolo F, Tiberi E, Barone G, Romagnoli C. Early weaning from incubator and early discharge of preterm infants: randomized clinical trial. Pediatrics. 2010 Sep;126(3):e651-6. doi: 10.1542/peds.2009-3005. Epub 2010 Aug 9. PMID 20696729
- [Background] Whyte RK. Neonatal management and safe discharge of late and moderate preterm infants. Semin Fetal Neonatal Med. 2012 Jun;17(3):153-8. doi: 10.1016/j.siny.2012.02.004. Epub 2012 Feb 24. PMID 22364676
- [Background] Heimler R, Sumners JE, Grausz JP, Kien CL, Glaspey JC. Thermal environment change in growing premature infants: effect on general somatic growth and subcutaneous fat accumulation. Pediatrics. 1981 Jul;68(1):82-6. PMID 7243513
- [Background] Barone G, Corsello M, Papacci P, Priolo F, Romagnoli C, Zecca E. Feasibility of transferring intensive cared preterm infants from incubator to open crib at 1600 grams. Ital J Pediatr. 2014 May 3;40:41. doi: 10.1186/1824-7288-40-41. PMID 24886971
- [Background] Schneiderman R, Kirkby S, Turenne W, Greenspan J. Incubator weaning in preterm infants and associated practice variation. J Perinatol. 2009 Aug;29(8):570-4. doi: 10.1038/jp.2009.54. Epub 2009 May 21. PMID 19461592